CLINICAL TRIAL: NCT02919904
Title: Feasibility of Using the ARESTM Device to Measure Sleep Parameters in Men With Asymptomatic Prostate Cancer Before as Well as at 3 and 6 Months After Starting Androgen Deprivation Therapy
Brief Title: Feasibility Study for the Assessment of Sleep Quality in Men With Prostate Cancer Starting ADT
Status: Completed | Type: Observational
Sponsor: Vancouver Prostate Centre (Other)
Responsible Party: Sponsor
Other Study IDs: Sleep Pilot
Record Dates: First submitted 2016-09-06; First posted 2016-09-29 (Estimated); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Prostatic Neoplasms; Sleep
Keywords: prostate cancer; sleep; androgen deprivation therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ARESTM — The ARESTM device is a commercial home sleep-testing device that can record the following parameters (for up to 7 continuous hours) when participants are asleep:
  * NREM and REM sleep frequency and duration
  * Duration and number of arousal
  * Blood oxygen saturation and pulse rate via a silicone-embedded optical sensor
  * Fluctuation in nasal airflow pressure via a nasal cannula and pressure transducer
  * Head movement actigraphy and flux in snoring as measures of sleep/wake patterns via two accelerometers and an acoustic microphone
  * Apnea/hypopnea index and respiratory disturbance index

SUMMARY:
The feasibility of using the Apnea Risk Evaluating System (ARESTM) device to take longitudinal measures of sleep parameters in asymptomatic men with prostate cancer who are about to initiate androgen deprivation therapy (ADT) will be evaluated. Study participants will complete serial questionnaires relating to sleep quality, hot flashes, and quality of life.

DETAILED DESCRIPTION:
The primary purpose of our study is to examine the feasibility of using the ARESTM device to measure sleep parameters of prostate cancer patients who are beginning ADT. Although some evidence links ADT to poor quality of sleep, no research has assessed the impact of ADT on most sleep parameters. We chose the ARESTM device for this study because the device can comprehensively measure sleep parameters. Furthermore, unlike polysomnography, the ARESTM device is easy to use and the measurements can be done at participants' home, without requiring them to adapt to a new sleeping location (e.g., sleep lab). ARESTM is a wireless device that is worn on the forehead during sleep to record physiological parameters. In addition, the feasibility of obtaining serial questionnaires from patients will be assessed. In this pilot study, the study investigators will attempt to make some preliminary correlations between sleep quality (as measured by ARESTM) with subjective sleep quality, morphometric measures, urinary symptoms, and hot flashes. Data collected from this study will help to determine the acceptability of and compliance with using the ARESTM device by this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed prostate cancer starting hormone therapy with or without concomitant radiation therapy for at least 6 months, or
2. Biochemical relapse of prostate cancer without metastatic symptoms (i.e. rising Prostate-specific antigen (PSA) after definitive therapy with no evidence of metastatic disease)*.
3. Serum testosterone in the hypogonadal range or above, but not at castrate levels.
4. About to start ADT with a Luteinizing Hormone-Releasing Hormone (LHRH) analogue for at least 6 months.
5. Fluent in English (able to read, write, and speak in English).
6. Provide written informed consent.
7. Patients with sleep apnea who do not depend on a CPAP (continuous positive airway pressure) machine to sleep may join the study.

   * Note: For participants who are having both hormone therapy and radiation, sleep parameters will only be measured before the participant starts radiation.

Exclusion Criteria:

1. Receiving antiandrogen monotherapy.
2. Previous history of sleep disorder (e.g., being treated for obstructive sleep apnea (and wear a CPAP machine), narcolepsy, parasomnia, circadian rhythm abnormalities).
3. Use of routine prescription or over the counter sleep medications (e.g., melatonin, zolpidem, suvorexant, eszopiclone, ramelteon, benzodiazepine, antihistamine).
4. Active medical problems that interfere with sleep (e.g. congestive heart failure).
5. Active medical problems that interfere with ARESTM reading or use of the device: deafness, blindness, severe arthritis, dementia, atrial fibrillation, tics or tremors of the head.
6. Use of supplemental oxygen at night.
7. Sensitivity of skin or scalp and/or open wounds on the forehead or scalp.
8. Allergic reactions to extended exposure to synthetics fabrics (e.g. polyester, rayon).
9. Upper respiratory infection or congestion.
10. Inability to sleep at least 5 hours per night or a total of 8 hours over two nights.
11. Inability to sleep with head reclined (less than 60 degree angle).
12. Head circumference less than 21 inches or greater than 25 inches.
13. Any reason that would prevent the participant from completing the study protocol or medical reason that would preclude them taking part.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 25 men starting androgen deprivation therapy for asymptomatic prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2015-07; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | up to 2 years
  Time taken to recruit men to this protocol will be measured

SECONDARY OUTCOMES:
Sleep quality parameters (composite outcome measure) | At baseline, 3 months and 6 months
  To measure parameters associated with sleep quality (non-rapid eye movement (NREM) & and rapid eye movement (REM), sleep frequency and duration, duration and number of awakenings, blood oxygen saturation and pulse rate, fluctuation in nasal airflow pressure, head movement actigraphy and flux in snoring as measures of sleep/wake patterns, apnea/hypopnea index and respiratory disturbance index).
Pittsburgh Sleep Quality Index (PSQI): subjective sleep quality | At baseline, 3 months and 6 months
  To assess subjective sleep quality. This questionnaire will be administered at the same time points as the sleep recordings are carried out.
Hot Flash Related Daily Interference Scale (HFRDIS) | At baseline, 3 months and 6 months
  To assess whether severe hot flash interferes with various daily activities. This questionnaire will be administered at the same time points as the sleep recordings are carried out.
Modified Expanded Prostate Cancer Index Composite (EPIC) | At baseline, 3 months and 6 months
  To assess study participant's urinary symptoms, frequency and how bothered they are with some ADT side effects (e.g. depression, fatigue, weight gain). This questionnaire will be administered at the same time points as the sleep recordings are carried out.

CONTACTS AND LOCATIONS:
Overall Officials: Larry Goldenberg, MD, Principal Investigator — University British Columbia
Locations (1):
- Vancouver Prostate Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No